CLINICAL TRIAL: NCT02160899
Title: A Randomized, Double Blind, Placebo-Controlled, Dose Titration, Phase 2 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ISIS 494372 Administered Subcutaneously to Patients With High Lipoprotein(a)
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ISIS-APO(a)Rx in Participants With High Lipoprotein(a)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 494372-CS3
Record Dates: First submitted 2014-06-05; First posted 2014-06-11 (Estimated); Results first posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Elevated Lipoprotein(a)
Keywords: High Lipoprotein(a)
MeSH Terms: interventions — ISIS-APO(a)Rx

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort A: Placebo (Placebo Comparator): Participants will receive placebo (normal saline) subcutaneously on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
  Interventions: Drug: Placebo
- Cohort A: ISIS-APO(a)Rx < 2000 mg (Experimental): Participants will receive ISIS-APO(a)Rx subcutaneously: 100 mg on Days 1, 8, 15, and 22; 200 mg on Days 29, 36, 43, and 50 unless down-titrated; and 300 mg on Days 57, 64, 71, and 78 unless down-titrated.
  Interventions: Drug: ISIS-APO(a)Rx
- Cohort A: ISIS-APO(a)Rx >= 2000 mg (Experimental): Participants will receive ISIS-APO(a)Rx subcutaneously: 100 mg on Days 1, 8, 15, and 22; 200 mg on Days 29, 36, 43, and 50 unless down-titrated; and 300 mg on Days 57, 64, 71, and 78 unless down-titrated.
  Interventions: Drug: ISIS-APO(a)Rx
- Cohort B: Placebo (Placebo Comparator): Participants will receive placebo (normal saline) subcutaneously on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
  Interventions: Drug: Placebo
- Cohort B: ISIS-APO(a)Rx < 2000 mg (Experimental): Participants will receive ISIS-APO(a)Rx subcutaneously: 100 mg on Days 1, 8, 15, and 22; 200 mg on Days 29, 36, 43, and 50 unless down-titrated; and 300 mg on Days 57, 64, 71, and 78 unless down-titrated.
  Interventions: Drug: ISIS-APO(a)Rx
- Cohort B: ISIS-APO(a)Rx >= 2000 mg (Experimental): Participants will receive ISIS-APO(a)Rx subcutaneously: 100 mg on Days 1, 8, 15, and 22; 200 mg on Days 29, 36, 43, and 50 unless down-titrated; and 300 mg on Days 57, 64, 71, and 78 unless down-titrated.
  Interventions: Drug: ISIS-APO(a)Rx

INTERVENTIONS:
Drug: ISIS-APO(a)Rx — ISIS-APO(a)Rx subcutaneously: 100 mg on Days 1, 8, 15, and 22; 200 mg on Days 29, 36, 43, and 50 unless down-titrated; and 300 mg on Days 57, 64, 71, and 78 unless down-titrated.
  Other Names: ISIS 494372
  Arms: Cohort A: ISIS-APO(a)Rx < 2000 mg; Cohort A: ISIS-APO(a)Rx >= 2000 mg; Cohort B: ISIS-APO(a)Rx < 2000 mg; Cohort B: ISIS-APO(a)Rx >= 2000 mg
Drug: Placebo — Normal saline as Placebo, subcutaneously on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
  Arms: Cohort A: Placebo; Cohort B: Placebo

SUMMARY:
The purpose is to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of ISIS-APO(a)Rx given to participants with high lipoprotein(a) for 12 weeks.

DETAILED DESCRIPTION:
Lipoprotein(a) [Lp(a)] is a genetic variant of low-density lipoprotein (LDL) in which the apolipoprotein B (apoB) -100 component of LDL is linked by a disulfide bond to apolipoprotein(a) [apo(a)], the distinct protein component of Lp(a) that is mainly responsible for its signature structural and functional properties. Lp(a) is now recognized as an important genetic risk factor for coronary artery disease, stroke and aortic stenosis.

The purpose of this study is to determine if ISIS-APO(a)Rx can reduce the production of apolipoprotein(a), or apo(a). This study will enroll 50 participants with Lipoprotein(a) ≥50 and <175 mg/dL and 10 participants with Lipoprotein(a) ≥175 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18-65 inclusive
* Females must be non-pregnant and non-lactating, and either surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or post-menopausal (defined as 12 months of spontaneous amenorrhea without an alternative medical cause and follicle-stimulating hormone (FSH) levels in the postmenopausal range for the laboratory involved)
* Males must be surgically sterile, abstinent or if engaged in sexual relations with a female of child-bearing potential, the participant must be using an acceptable contraceptive method from the time of signing the informed consent form until at least 16 weeks after the last dose of Study Drug
* Body mass index (BMI) ≤40 kg/m2
* Lipoprotein(a) ≥50 and <175 mg/dL at time of screening (Cohort A)
* Lipoprotein(a) ≥175 mg/dL at time of screening (Cohort B)

Exclusion Criteria:

* Clinically significant abnormalities in medical history (e.g., documented previous myocardial infarction, percutaneous coronary intervention (PCI), or major surgery within 3 months of screening, planned surgery that would occur during the study) or physical examination at screening
* Clinically significant abnormalities in screening laboratory values that would render a participant unsuitable for inclusion
* Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
* Known history or positive test for human immunodeficiency virus (HIV), hepatitis C, or chronic hepatitis B
* Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated
* History of bleeding diathesis or coagulopathy
* Recent history of, or current drug or alcohol abuse
* Participant with Lp(a) ≥50 and <175 mg/dL may not receive concomitant niacin therapy during the period 8 weeks prior to screening through the end of the Post-Treatment Evaluation Period
* Use of statins, ezetimibe or fibrates unless on a stable regimen for at least 8 weeks prior to dosing and will remain on a stable regimen for the duration of the study
* Use of lipid or Lp(a)-specific apheresis within 4 weeks prior to Screening through the end of the Post-Treatment Evaluation Period
* Use of concomitant drugs (including herbal or over-the-counter (OTC) medications other than ibuprofen, Benadryl or topical steroids) unless authorized by the Sponsor Medical Monitor
* Blood donation of 50-499 mL within 30 days of screening or of >499 mL within 8 weeks of screening
* Have any other conditions, which, in the opinion of the Investigator would make the participant unsuitable for inclusion, or could interfere with the participant participating in or completing the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Canada (2):
  - Chicoutimi Hospital, Chicoutimi, Quebec
  - Clinique des Maladies Lipidiques de Quebec Inc., Québec
- Herlev University Hospital, Herlev, Denmark
- Germany (3):
  - Charite - University Hospital Berlin - Campus Virchow - Hospital, Berlin
  - Uniklinik Koeln, Zentrum fuer Endokrinologie, Diabetologie und Praeventivmedizin (ZEDP), Cologne
  - Otto-von Guericke Universitaet, Uniklinik Magdeburg, Magdeburg
- Netherlands (4):
  - University of Amsterdam - Dept. of Vascular Medicine F4-109, Amsterdam
  - Academic Hospital Maastricht, Maastricht
  - Sint Franciscus Gasthuis, Rotterdam
  - University Medical Center Utrecht, Utrecht
- United Kingdom (3):
  - Heart of England NHS Foundation Trust, Birmingham
  - Barlow Medical Centre, Manchester
  - Newcastle Upon Tyne Hospitals, Newcastle upon Tyne

REFERENCES:
- [Derived] Viney NJ, van Capelleveen JC, Geary RS, Xia S, Tami JA, Yu RZ, Marcovina SM, Hughes SG, Graham MJ, Crooke RM, Crooke ST, Witztum JL, Stroes ES, Tsimikas S. Antisense oligonucleotides targeting apolipoprotein(a) in people with raised lipoprotein(a): two randomised, double-blind, placebo-controlled, dose-ranging trials. Lancet. 2016 Nov 5;388(10057):2239-2253. doi: 10.1016/S0140-6736(16)31009-1. Epub 2016 Sep 21. PMID 27665230
- [Derived] Tragante V, Asselbergs FW, Swerdlow DI, Palmer TM, Moore JH, de Bakker PIW, Keating BJ, Holmes MV. Harnessing publicly available genetic data to prioritize lipid modifying therapeutic targets for prevention of coronary heart disease based on dysglycemic risk. Hum Genet. 2016 May;135(5):453-467. doi: 10.1007/s00439-016-1647-9. Epub 2016 Mar 5. PMID 26946290

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 51 participants were enrolled in Cohort A and 13 participants were enrolled in Cohort B.
Pre-assignment Details: A total of 86 participants were screened for the study and 64 participants were randomized into Cohort A and Cohort B and received study treatment. Two participants in Cohort B did not complete the study treatment but completed the post-treatment follow-up.
Groups:
- Cohort A: Placebo; Cohort B: Placebo: Participants received placebo (normal saline) subcutaneously on Days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
- Cohort A: ISIS-APO(a)Rx < 2000 mg; Cohort A: ISIS-APO(a)Rx >= 2000 mg; Cohort B: ISIS-APO(a)Rx < 2000 mg; Cohort B: ISIS-APO(a)Rx >= 2000 mg: Participants received ISIS-APO(a)Rx subcutaneously: 100 mg on Days 1, 8, 15, and 22; 200 mg on Days 29, 36, 43, and 50 unless down-titrated; and 300 mg on Days 57, 64, 71, and 78 unless down-titrated.
Period: Overall Study
Arm/Group | Cohort A: Placebo | Cohort A: ISIS-APO(a)Rx < 2000 mg | Cohort A: ISIS-APO(a)Rx >= 2000 mg | Cohort B: Placebo | Cohort B: ISIS-APO(a)Rx < 2000 mg | Cohort B: ISIS-APO(a)Rx >= 2000 mg
Started | 26 | 4 | 21 | 3 | 2 | 8
Completed | 26 | 3 | 21 | 2 | 0 | 8
Not Completed | 0 | 1 | 0 | 1 | 2 | 0
Not completed — Adverse Event or Serious Adverse Event | 0 | 1 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Set included all randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Placebo | Cohort A: ISIS-APO(a)Rx < 2000 mg | Cohort A: ISIS-APO(a)Rx >= 2000 mg | Cohort B: Placebo | Cohort B: ISIS-APO(a)Rx < 2000 mg | Cohort B: ISIS-APO(a)Rx >= 2000 mg | Total
Number analyzed (Participants) | 26 | 4 | 21 | 3 | 2 | 8 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10) | 50 (9) | 56 (6) | 62 (8) | 45 (11) | 61 (8) | 55 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 12 | 3 | 2 | 6 | 31
  Male | 20 | 2 | 9 | 0 | 0 | 2 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 4 | 21 | 3 | 2 | 8 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 25 | 4 | 20 | 3 | 2 | 8 | 62
  Black | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Other Race | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lipoprotein Lp(a) Plasma Concentration at Day 85/Day 99
Description: Data are reported for evaluable participants.
Time Frame: Day 85/Day 99
Population: The Per-Protocol Set included the subset of the Full Analysis Set who received at least 9 doses of Study Drug within the 12-week treatment period and who had no significant protocol deviations that would have been expected to affect efficacy assessments. Day 85/Day 99 result is defined as the result at Day 85 or Day 99.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort A: Placebo | Cohort A: ISIS-APO(a)Rx < 2000 mg | Cohort A: ISIS-APO(a)Rx >= 2000 mg | Cohort B: Placebo | Cohort B: ISIS-APO(a)Rx < 2000 mg | Cohort B: ISIS-APO(a)Rx >= 2000 mg
Number analyzed (Participants) | 26 | 3 | 21 | 2 | 0 | 8
percent change | -3.7 (13.7) | -44.5 (13.1) | -70.0 (19.6) | -5.6 (3.9) |  | -71.6 (13.0)
Statistical Analysis 1: Comparison: Cohort A: Placebo vs Cohort A: ISIS-APO(a)Rx < 2000 mg; Test type: Superiority; p < .001, ANOVA
Statistical Analysis 2: Comparison: Cohort A: Placebo vs Cohort A: ISIS-APO(a)Rx >= 2000 mg; Test type: Superiority; p < .001, ANOVA
Statistical Analysis 3: Comparison: Cohort B: Placebo vs Cohort B: ISIS-APO(a)Rx >= 2000 mg; Test type: Superiority; p = 0.044, Exact Wilcoxon Rank Sum Test

2. Primary Outcome: Number of Participants With at Least One Treatment-emergent Adverse Event (TEAE)
Description: An adverse event is any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.
Time Frame: Up to approximately 32 weeks
Population: The Safety Set included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Placebo | Cohort A: ISIS-APO(a)Rx < 2000 mg | Cohort A: ISIS-APO(a)Rx >= 2000 mg | Cohort B: Placebo | Cohort B: ISIS-APO(a)Rx < 2000 mg | Cohort B: ISIS-APO(a)Rx >= 2000 mg
Number analyzed (Participants) | 26 | 4 | 21 | 3 | 2 | 8
Participants | 23 | 4 | 21 | 2 | 2 | 8

ADVERSE EVENTS:
Time Frame: Up to approximately 32 weeks
Description: The Safety Set included all randomized participants who received at least one dose of study drug.
Arm/Group | Cohort A: Placebo | Cohort A: ISIS-APO(a)Rx < 2000 mg | Cohort A: ISIS-APO(a)Rx >= 2000 mg | Cohort B: Placebo | Cohort B: ISIS-APO(a)Rx < 2000 mg | Cohort B: ISIS-APO(a)Rx >= 2000 mg
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/4 | 0/21 | 0/3 | 0/2 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/26 | 2/4 | 0/21 | 1/3 | 0/2 | 0/8
Other Adverse Events (participants affected / at risk) | 23/26 | 3/4 | 21/21 | 2/3 | 2/2 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Placebo (N=26) | Cohort A: ISIS-APO(a)Rx < 2000 mg (N=4) | Cohort A: ISIS-APO(a)Rx >= 2000 mg (N=21) | Cohort B: Placebo (N=3) | Cohort B: ISIS-APO(a)Rx < 2000 mg (N=2) | Cohort B: ISIS-APO(a)Rx >= 2000 mg (N=8)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Placebo (N=26) | Cohort A: ISIS-APO(a)Rx < 2000 mg (N=4) | Cohort A: ISIS-APO(a)Rx >= 2000 mg (N=21) | Cohort B: Placebo (N=3) | Cohort B: ISIS-APO(a)Rx < 2000 mg (N=2) | Cohort B: ISIS-APO(a)Rx >= 2000 mg (N=8)
Injection site erythema (General disorders) | 0 | 3 | 16 | 0 | 2 | 6
Injection site pain (General disorders) | 2 | 1 | 12 | 0 | 2 | 2
Injection site induration (General disorders) | 0 | 3 | 8 | 0 | 0 | 4
Injection site swelling (General disorders) | 0 | 1 | 10 | 0 | 1 | 3
Injection site warmth (General disorders) | 0 | 0 | 2 | 0 | 1 | 3
Fatigue (General disorders) | 3 | 2 | 3 | 0 | 0 | 3
Injection site pruritus (General disorders) | 0 | 2 | 8 | 0 | 0 | 3
Injection site reaction (General disorders) | 1 | 0 | 7 | 0 | 1 | 1
Injection site hyperaesthesia (General disorders) | 0 | 0 | 2 | 0 | 0 | 3
Injection site discolouration (General disorders) | 0 | 0 | 5 | 0 | 0 | 2
Chills (General disorders) | 1 | 2 | 3 | 1 | 0 | 1
Malaise (General disorders) | 3 | 0 | 4 | 0 | 0 | 2
Injection site haematoma (General disorders) | 2 | 0 | 3 | 0 | 0 | 1
Injection site bruising (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Injection site urticaria (General disorders) | 0 | 0 | 3 | 0 | 0 | 2
Asthenia (General disorders) | 2 | 1 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 1 | 0 | 2
Hyperthermia (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 0 | 0 | 2
Injection site oedema (General disorders) | 0 | 0 | 2 | 0 | 0 | 1
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0
Injection site pallor (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 3 | 0 | 0 | 0 | 0 | 0
Injection site paraesthesia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 9 | 0 | 8 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 3 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0
Bacteriuria (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 6 | 1 | 10 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 3 | 0 | 4 | 0 | 0 | 2
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 3 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 2 | 2 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erythema annulare (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
General physical condition abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes